CLINICAL TRIAL: NCT03672461
Title: A Randomized Controlled Trial of a Group-Based Therapeutic Yoga Intervention for Urinary Incontinence in Ambulatory Older Women
Brief Title: A Group-Based Therapeutic Yoga Intervention for Urinary Incontinence in Ambulatory Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P0529491; R01DK116712-01A1 (NIH)
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Stress Incontinence, Female; Stress Incontinence, Urinary; Stress Incontinence; Urge Incontinence; Urinary Incontinence, Stress; Urinary Stress Incontinence; Urgency Urinary
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Practice Program (Experimental): The 3-month yoga intervention will provide instruction and practice in a variety of yoga postures and techniques that have been selected by the study yoga expert consultants for their potential to improve bladder control and safety and feasibility for the target population. The study will feature a therapeutic program based primarily on Iyengar yoga, a form of Hatha yoga that is known for its potential therapeutic applications.
  Interventions: Other: Yoga Practice Program
- Physical Conditioning Program (Active Comparator): The 3-month muscle stretching/strengthening intervention program (also referred to as the "physical conditioning" program) has been designed by the study physical therapist consultants. Similar to postures in the yoga intervention program, the exercises in the stretching/strengthening program have been selected for their potential to be performed safely by women across a range of ages and flexibility levels.
  Interventions: Other: Physical Conditioning Program

INTERVENTIONS:
Other: Yoga Practice Program — The 3-month yoga intervention will provide instruction and practice in a variety of yoga postures and techniques that have been selected by the study yoga expert consultants for their potential to improve bladder control and safety and feasibility for the target population.
  Arms: Yoga Practice Program
Other: Physical Conditioning Program — The 3-month muscle stretching/strengthening intervention program (also referred to as the "physical conditioning" program) has been designed by the study physical therapist consultants.
  Arms: Physical Conditioning Program

SUMMARY:
The investigators will conduct a randomized controlled trial to evaluate the efficacy of a group-based yoga intervention to decrease the frequency and impact of urinary incontinence in ambulatory middle-aged and older women and explore potential mediators of improvement in outcomes. Women aged 45 years and older who report daily or more frequent stress-, urgency-, or mixed-type incontinence, are not already engaged in formal yoga or muscle stretching/strengthening programs, are willing to temporarily forgo other clinical treatments for incontinence, are able to walk to and use the bathroom without assistance, and meet other eligibility criteria will be recruited from multiple locations surrounding the San Francisco Bay area.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45 years or older who report urinary incontinence starting at least 3 months prior to screening
* Self-report an average of at least one incontinence episode per day on a validated voiding diary
* Self-report urgency-predominant (i.e., at least half of incontinence episodes being urgency-type), stress-predominant (i.e., at least half of episodes being stress-type), or mixed-type (i.e., an equal number of stress- and urgency-type episodes) incontinence on the screening voiding diary
* Willing to refrain from initiating medical treatments that may affect their incontinence or voiding pattern during the study intervention period

Exclusion Criteria:

* Current participation in organized yoga classes or workshops, or any prior organized yoga training directed specifically at improving incontinence
* Current participation in organized physical conditioning classes involving muscle strengthening exercises (e.g., Pilates)
* Current urinary tract infection or hematuria detected by urinalysis at screening visit (women can re-present after evaluation and treatment through their usual care)
* Currently pregnant (by self-report or screening urine pregnancy test), gave birth within the past 3 months, or planning pregnancy during the study period
* Report use of medical devices (i.e. pessary) for incontinence within the past month (participants may stop use of device and re-present for study)
* Report use of bladder botox, electrostimulation, formal bladder training, or formal pelvic floor exercise training (with certified practitioners) in the past 3 months
* Report any history of prior anti-incontinence or urethral surgery (not including urethral dilation), pelvic cancer, or pelvic irradiation
* Report other surgery to the pelvis (hysterectomy, oophorectomy, vaginal surgery, bladder surgery, colon surgery) within the past 3 months
* Unable to walk 2 blocks on level ground without assistance (functional capacity < 4 metabolic equivalents)
* Unable to get up from a supine to a standing position without assistance (assessed during the screening visit)
* Report history of interstitial cystitis, bladder or rectal fistula, or congenital defect causing urinary incontinence
* Report incontinence caused by a major neurologic conditions such as multiple sclerosis, spinal cord injury, or Parkinson's disease
* Report use of medications with strong effects on urination (anticholinergic bladder medications, beta-3 agonists, tricyclic antidepressants, mirabegron, loop diuretics) within the past month
* Report starting, stopping, or changing the dose of a medication with the potential to affect anxiety or depression symptoms (i.e., selective serotonin reuptake inhibitors, anxiolytics/sedatives, antipsychotics) within the past 1 month, or plans to start, stop, or change to dose of such a medication during the study period
* Participation in another research study that involves investigational drugs or devices that could potentially confound the results of this study
* Unable to understand study procedures, complete study interviews, or and provide informed consent in English
* Report conditions that, in the judgment of the investigators, render potential participants unlikely to follow the protocol, including plans to move, substance abuse, significant psychiatric problems, or dementia

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Huang, MS, MAS, MPhil, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hough E, Goldstein LA, Subak LL, Chesney MA, Schembri M, Raghunathan H, Balys Pawlowsky S, Huang AJ. Effects of Hatha Yoga vs Physical Conditioning on Sleep in Women With Urinary Incontinence: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2546499. doi: 10.1001/jamanetworkopen.2025.46499. PMID 41359336
- [Derived] Huang AJ, Chesney M, Schembri M, Raghunathan H, Vittinghoff E, Mendes WB, Pawlowsky S, Subak LL. Efficacy of a Therapeutic Pelvic Yoga Program Versus a Physical Conditioning Program on Urinary Incontinence in Women : A Randomized Trial. Ann Intern Med. 2024 Oct;177(10):1339-1349. doi: 10.7326/M23-3051. Epub 2024 Aug 27. PMID 39186785
- [Derived] Huang AJ, Chesney MA, Schembri M, Pawlowsky S, Nicosia F, Subak LL. Rapid Conversion of a Group-Based Yoga Trial for Diverse Older Women to Home-Based Telehealth: Lessons Learned Using Zoom to Deliver Movement-Based Interventions. J Integr Complement Med. 2022 Feb;28(2):188-192. doi: 10.1089/jicm.2021.0268. Epub 2022 Jan 10. PMID 35167358

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Started | 121 | 119
Completed | 101 | 109
Not Completed | 20 | 10
Not completed — COVID Related | 4 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Serious Adverse Event | 0 | 1
Not completed — Too Busy | 3 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Family | 2 | 2
Not completed — No remote technology access | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Cannot tolerate intervention | 1 | 0
Not completed — Incomplete outcome data | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga Practice Program | Physical Conditioning Program | Total
Number analyzed (Participants) | 121 | 119 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.7) | 61.4 (8.8) | 62.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 119 | 240
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 83 | 77 | 160
  Black | 7 | 12 | 19
  Hispanic | 21 | 11 | 32
  Asian | 20 | 20 | 40
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  American Indian | 0 | 0 | 0
  Other | 0 | 1 | 1
  More than one race | 11 | 9 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 121 | 119 | 240
Total Urinary Incontinence Episodes [Mean (Standard Deviation); unit: episodes per day] | 3.6 (2.5) | 3.2 (1.9) | 3.4 (2.2)
Stress-Type Urinary Incontinence Episodes [Mean (Standard Deviation); unit: episodes per day] | 1.4 (1.8) | 1.4 (1.5) | 1.4 (1.6)
Urgency-Type Urinary Incontinence Episodes [Mean (Standard Deviation); unit: episodes per day] | 2.1 (2.2) | 1.7 (1.4) | 1.9 (1.9)
Incontinence Impact Questionnaire (IIQ) [Mean (Standard Deviation); unit: units on a scale] — Range 0-400, higher score indicates lower quality of life.
  units on a scale | 100.4 (78.9) | 101.6 (66.4) | 101.0 (72.7)
Urogenital distress inventory-6 score (UDI) [Mean (Standard Deviation); unit: units on a scale] — Range 0-100, higher score indicates lower quality of life.
  units on a scale | 39.1 (19.1) | 38.5 (19.4) | 38.8 (19.2)
Patient Perception of Bladder Condition (PPBC) [Mean (Standard Deviation); unit: units on a scale] — Range 1-6, higher score indicates lower quality of life.
  units on a scale | 3.3 (1.0) | 3.4 (1.0) | 3.4 (1.0)
Center for Epidemiologic Studies Depression Scale (CES-D) [Mean (Standard Deviation); unit: units on a scale] — Range 0-60, higher score indicates lower quality of life.
  units on a scale | 10.1 (8.8) | 10.0 (8.1) | 10.0 (8.4)
State/Trait Anxiety Inventory (STAI)--Trait [Mean (Standard Deviation); unit: units on a scale] — Range 20-80, higher score indicates lower quality of life.
  units on a scale | 36.1 (11.2) | 36.1 (10.5) | 36.1 (10.9)
Hospital Anxiety & Depression (HADS)--Anxiety score [Mean (Standard Deviation); unit: units on a scale] — Range 0-21, higher score indicates lower quality of life.
  units on a scale | 5.3 (3.8) | 5.2 (3.7) | 5.3 (3.8)
Perceived Stress Scale (PSS) score [Mean (Standard Deviation); unit: units on a scale] — Range 0-40, higher score indicates lower quality of life.
  units on a scale | 13.0 (7.2) | 13.3 (6.8) | 13.2 (7.0)
PROMIS Physical 8B, T-Score [Mean (Standard Deviation); unit: T-Score] — (mean 50, Std Dev 10) no widely accepted thresholds have been published. Range 20.9-59.7, Higher score indicates better quality of life.
  T-Score | 51.0 (6.2) | 51.3 (6.8) | 51.2 (6.5)
One-legged Balance Test [Mean (Standard Deviation); unit: seconds] — Range 0-30 seconds
  seconds | 24.4 (9.9) | 25.5 (8.7) | 24.9 (9.4)
Chair Stands (in 30 seconds) [Mean (Standard Deviation); unit: chair stands] | 12.6 (3.9) | 13.1 (4.2) | 12.9 (4.1)
2-Minute Step Test [Mean (Standard Deviation); unit: steps] | 85.9 (22.8) | 88.5 (26.1) | 87.2 (24.5)
Wake after sleep onset [Mean (Standard Deviation); unit: minutes] | 24.4 (29.2) | 25.2 (25.6) | 24.8 (27.4)
Total sleep time [Mean (Standard Deviation); unit: Hours] | 7.1 (1.2) | 7.0 (1.0) | 7.0 (1.1)
Pittsburgh Sleep Quality Index (PSQI) total score [Mean (Standard Deviation); unit: units on a scale] — Range 0-21, higher score indicates lower quality of life.
  units on a scale | 6.2 (3.1) | 6.6 (3.1) | 6.4 (3.1)
Pelvic Organ Prolapse/Incontinence Sexual Questionnaire IUGA-Revised (PISQ-IR) [Mean (Standard Deviation); unit: units on a scale] — Range for each subscale 0-100. Higher score indicates higher quality of life. Population: The domains are specific to two distinct groups: Sexually active (SA) and Not Sexually Active (NSA). 4 NSA variables: Domains relevant only to participants that are not sexually active. 6 SA variables: Domains relevant only to sexually active participants. Additional missingness is due to not having a partner (SA), or to survey or item non-response.
  units on a scale
    PISQ-IR Sexually Inactive, Condition Impact on Sexual Quality: number analyzed (Participants) | 55 | 50 | 105
    PISQ-IR Sexually Inactive, Condition Impact on Sexual Quality | 21.6 (26.9) | 13.6 (21.6) | 17.8 (24.7)
    PISQ-IR Sexually Inactive, Condition Specific Reason for Not Being Active: number analyzed (Participants) | 54 | 47 | 101
    PISQ-IR Sexually Inactive, Condition Specific Reason for Not Being Active | 24.8 (21.9) | 19.6 (22.2) | 22.4 (22.1)
    PISQ-IR Sexually Inactive, Global Quality: number analyzed (Participants) | 55 | 50 | 105
    PISQ-IR Sexually Inactive, Global Quality | 48.6 (29.6) | 49.6 (32.5) | 49.1 (30.9)
    PISQ-IR Sexually Inactive, Partner-Related Reasons for Not Being Active: number analyzed (Participants) | 54 | 50 | 104
    PISQ-IR Sexually Inactive, Partner-Related Reasons for Not Being Active | 56.8 (26.0) | 60.0 (23.6) | 58.3 (24.8)
    PISQ-IR Sexually Active, Assessment of Arousal, Orgasm: number analyzed (Participants) | 61 | 68 | 129
    PISQ-IR Sexually Active, Assessment of Arousal, Orgasm | 63.2 (12.8) | 63.3 (17.3) | 63.3 (15.3)
    PISQ-IR Sexually Active, Condition-specific Impact on Sexual Quality: number analyzed (Participants) | 61 | 68 | 129
    PISQ-IR Sexually Active, Condition-specific Impact on Sexual Quality | 81.4 (23.4) | 79.4 (20.3) | 80.4 (21.8)
    PISQ-IR Sexually Active, Condition-specifc Impacts on Activity: number analyzed (Participants) | 61 | 68 | 129
    PISQ-IR Sexually Active, Condition-specifc Impacts on Activity | 86.2 (13.9) | 87.0 (12.8) | 86.6 (13.3)
    PISQ-IR Sexually Active, Assessment of Desire: number analyzed (Participants) | 61 | 68 | 129
    PISQ-IR Sexually Active, Assessment of Desire | 48.6 (18.1) | 50.1 (18.3) | 49.4 (18.2)
    PISQ-IR Sexually Active, Global Quality: number analyzed (Participants) | 61 | 68 | 129
    PISQ-IR Sexually Active, Global Quality | 62.2 (28.3) | 64.0 (28.1) | 63.2 (28.1)
    PISQ-IR Sexually Active Interest, Assessment of Partner Related Impacts: number analyzed (Participants) | 54 | 54 | 108
    PISQ-IR Sexually Active Interest, Assessment of Partner Related Impacts | 77.2 (17.1) | 77.0 (19.0) | 77.1 (18.0)
    PISQ-IR Sexually Active Interest, Summary Score: number analyzed (Participants) | 61 | 68 | 129
    PISQ-IR Sexually Active Interest, Summary Score | 68.8 (13.2) | 68.9 (13.8) | 68.9 (13.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Urinary Incontinence Episodes
Description: Change was calculated as the followup value minus the baseline value. Values are model-generated Least Square Means for combined 6 and 12 week time points.
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: episodes per day
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 106 | 113
episodes per day | -1.99 [-2.21 to -1.77] | -1.7 [-1.91 to -1.49]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Null Hypothesis: Yoga is not associated with improvement in change from baseline in Total Urinary Incontinence Episodes; Test type: Superiority; p = 0.056, Mixed Models Analysis; adjusted for baseline value. Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.29, 95% CI 2-sided [-0.01 to 0.6]

2. Secondary Outcome: Change From Baseline in Stress-Type Urinary Incontinence Episodes
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: episodes per day
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 106 | 113
episodes per day | -0.8 [-0.93 to -0.67] | -0.77 [-0.9 to -0.65]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.757, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.03, 95% CI 2-sided [-0.15 to 0.2]

3. Secondary Outcome: Change From Baseline in Urgency-Type Urinary Incontinence Episodes
Description: Change was calculated as the follow-up value minus the baseline value. Values are model-generated Least Square Means for combined 6 and 12 week time points
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: episodes per day
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 106 | 113
episodes per day | -1.12 [-1.28 to -0.96] | -0.9 [-1.06 to -0.74]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.048, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.22, 95% CI 2-sided [0 to 0.45]

4. Secondary Outcome: Change From Baseline in Incontinence Impact Questionnaire (IIQ)
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points Range 0-400, Higher score indicates lower quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 107 | 112
units on a scale | -31.3 [-41.6 to -20.9] | -30.4 [-40.7 to -20.2]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.911, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.82, 95% CI 2-sided [-13.6 to 15.23]

5. Secondary Outcome: Change From Baseline in Urogenital Distress Inventory-6 Score (UDI)
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points Range 0-100, Higher score indicates lower quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 108 | 112
units on a scale | -14.9 [-17 to -12.7] | -11.7 [-13.9 to -9.59]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.041, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 3.13, 95% CI 2-sided [0.13 to 6.13]

6. Secondary Outcome: Change From Baseline in Patient Perception of Bladder Condition (PPBC)
Description: Change was calculated as the follow-up value minus the baseline value. Values are model-generated Least Square Means for combined 6 and 12 week time points Range 1-6, Higher score indicates lower quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 107 | 112
units on a scale | -0.59 [-0.75 to -0.42] | -0.52 [-0.69 to -0.36]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.564, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.07, 95% CI 2-sided [-0.16 to 0.3]

7. Secondary Outcome: Change From Baseline in Center for Epidemiologic Studies Depression Scale (CES-D)
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points Range 0-60, Higher score indicates lower quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 107 | 112
units on a scale | -0.82 [-2.25 to 0.6] | -0.52 [-1.93 to 0.9]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.764, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.3, 95% CI 2-sided [-1.69 to 2.3]

8. Secondary Outcome: Change From Baseline in State/Trait Anxiety Inventory (STAI)--Trait
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points Range 20-80, Higher score indicates lower quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 107 | 112
units on a scale | -1.22 [-2.41 to -0.03] | -1.34 [-2.52 to -0.17]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.883, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -0.12, 95% CI 2-sided [-1.78 to 1.53]

9. Secondary Outcome: Change From Baseline in Hospital Anxiety & Depression (HADS)--Anxiety Score
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points Range 0-21, Higher score indicates lower quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 107 | 111
units on a scale | -0.21 [-0.72 to 0.3] | -0.33 [-0.83 to 0.18]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.753, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -0.11, 95% CI 2-sided [-0.83 to 0.6]

10. Secondary Outcome: Change From Baseline in Perceived Stress Scale (PSS) Score
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points Range 0-40, Higher score indicates lower quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 106 | 112
units on a scale | -0.44 [-1.41 to 0.52] | -0.72 [-1.68 to 0.24]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.685, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -0.28, 95% CI 2-sided [-1.63 to 1.07]

11. Secondary Outcome: Change From Baseline in PROMIS Physical Function Short Form 8B, T-Score
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points (Mean 50, Std Dev 10) no widely accepted thresholds have been published. Higher score indicates better quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 106 | 109
T-score | -0.2 [-1.05 to 0.65] | 0.04 [-0.81 to 0.89]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.691, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.24, 95% CI 2-sided [-0.95 to 1.43]

12. Secondary Outcome: Change From Baseline in One-legged Balance Test (Winsorized)
Description: Change was calculated as the followup value minus the baseline value. Change values were Winsorized at the 1st and 99th percentile. Values are model generated Least Square Means for combined 6 and 12 week time points. Higher score indicates better quality of life.
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 107 | 110
seconds | 1.34 [0.52 to 2.16] | 1.53 [0.72 to 2.35]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.743, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.19, 95% CI 2-sided [-0.95 to 1.34]

13. Secondary Outcome: Change From Baseline in Chair Stands (in 30 Seconds)
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points Higher score indicates better quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: chair stands
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 105 | 106
chair stands | 1 [0.32 to 1.68] | 1.98 [1.3 to 2.66]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.043, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.98, 95% CI 2-sided [0.03 to 1.93]

14. Secondary Outcome: Change From Baseline in 2-Minute Step Test
Description: as for outcome 13
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: steps
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 104 | 109
steps | 8.05 [4.58 to 11.51] | 9.03 [5.59 to 12.48]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.689, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.99, 95% CI 2-sided [-3.87 to 5.84]

15. Secondary Outcome: Change From Baseline in Wake After Sleep Onset (Winsorized)
Description: Change was calculated as the follow-up value minus the baseline value. Change values were Winsorized at the 1st and 99th percentile. Values are model generated Least Square Means for combined 6 and 12 week time points.
  Higher score indicates lower quality of life.
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 104 | 108
minutes | -3.55 [-7.96 to 0.85] | -6.96 [-11.3 to -2.61]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.276, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -3.4, 95% CI 2-sided [-9.54 to 2.74]

16. Secondary Outcome: Change From Baseline in Total Sleep Time
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points.
  Higher score indicates better quality of life.
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: hours
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 104 | 109
hours | 0 [-0.18 to 0.17] | 0.09 [-0.08 to 0.27]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.448, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 0.1, 95% CI 2-sided [-0.15 to 0.34]

17. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) Total Score
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points.
  Range of 0-21, higher score indicates lower quality of life.
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Number of participants with outcomes data
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 108 | 112
units on a scale | -0.37 [-0.78 to 0.04] | -0.66 [-1.07 to -0.25]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.319, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -0.29, 95% CI 2-sided [-0.86 to 0.28]

18. Secondary Outcome: Change From Baseline in Pelvic Organ Prolapse/Incontinence Sexual Questionnaire IUGA-Revised (PISQ-IR)--Sexually Inactive, Condition Impact on Sexual Quality
Description: Change was calculated as the followup value minus the baseline value. Values are model generated Least Square Means for combined 6 and 12 week time points Range of 0-100, higher score indicates better quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Domains relevant only to participants that are not sexually active. Additional missingness is due to not having a partner (SA), or to survey or item non-response.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 38 | 44
units on a scale | -5.04 [-10.7 to 0.58] | -3.83 [-8.84 to 1.19]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.747, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 1.21, 95% CI 2-sided [-6.25 to 8.67]

19. Secondary Outcome: Change From Baseline in Pelvic Organ Prolapse/Incontinence Sexual Questionnaire IUGA-Revised (PISQ-IR)--Sexually Inactive, Condition Specific Reason for Not Being Active
Description: Change was calculated as the follow-up value minus the baseline value. Values are model-generated Least Square Means for combined 6 and 12 week time points Range of 0-100, higher score indicates better quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: as for outcome 18
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 38 | 40
units on a scale | -1 [-6.52 to 4.52] | -3.76 [-8.86 to 1.35]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.459, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -2.76, 95% CI 2-sided [-10.2 to 4.65]

20. Secondary Outcome: Change From Baseline in Pelvic Organ Prolapse/Incontinence Sexual Questionnaire IUGA-Revised (PISQ-IR)--Sexually Inactive, Global Quality
Description: as for outcome 18
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: as for outcome 18
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 38 | 43
units on a scale | 1.3 [-3.67 to 6.27] | -0.67 [-5.27 to 3.93]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.556, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -2., 95% CI 2-sided [-10.2 to 4.65]

21. Secondary Outcome: Change From Baseline in Pelvic Organ Prolapse/Incontinence Sexual Questionnaire IUGA-Revised (PISQ-IR)--Sexually Inactive, Partner Related Reasons for Not Being Active
Description: as for outcome 18
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: as for outcome 18
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 38 | 43
units on a scale | 1.73 [-5.52 to 8.98] | -1.52 [-8.52 to 5.47]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.516, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -3.26, 95% CI 2-sided [-13.2 to 6.7]

22. Secondary Outcome: Change From Baseline in Pelvic Organ Prolapse/Incontinence Sexual Questionnaire IUGA-Revised (PISQ-IR)--Sexually Active, Assessment of Arousal, Orgasm
Description: as for outcome 18
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Domain is relevant only the sexually active participants
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 57 | 61
units on a scale | 0.83 [-1.54 to 3.2] | -1.55 [-3.85 to 0.75]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.154, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -2.38, 95% CI 2-sided [-5.68 to 0.91]

23. Secondary Outcome: Change From Baseline in Pelvic Organ Prolapse/Incontinence Sexual Questionnaire IUGA-Revised (PISQ-IR)--Sexually Active, Condition-specific Impact on Sexual Quality
Description: as for outcome 18
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Domain is relevant only the sexually active participants. Additional missingness is due to not having a partner (SA), or to survey or item non-response.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 56 | 62
units on a scale | 2.84 [-0.74 to 6.42] | 0.62 [-2.81 to 4.04]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.375, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -2.22, 95% CI 2-sided [-7.17 to 2.72]

24. Secondary Outcome: Change From Baseline in Pelvic Organ Prolapse/Incontinence Sexual Questionnaire IUGA-Revised (PISQ-IR)--Sexually Active, Condition-specifc Impacts on Activity
Description: as for outcome 18
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Domain is relevant only the sexually active participants
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 57 | 61
units on a scale | 3.7 [1.36 to 6.05] | 1.95 [1.95 to 4.22]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.287, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, with unstructured variance co-variance matrix; Model based LS mean difference = -1.75, 95% CI 2-sided [-5 to 1.5]

25. Secondary Outcome: Change From Baseline in Pelvic Organ Prolapse/Incontinence Sexual Questionnaire IUGA-Revised (PISQ-IR)--Sexually Active Interest, Summary Score
Description: as for outcome 19
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Domain is relevant only the sexually active participants
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 57 | 61
units on a scale | 1.47 [-0.12 to 3.07] | -0.16 [-1.71 to 1.39]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.147, Mixed Models Analysis — adjusted for baseline value Repeated measures mixed models, with unstructured variance co-variance matrix; Model based LS mean difference = -1.63, 95% CI 2-sided [-3.85 to 0.58]

26. Secondary Outcome: Change From Baseline in Pelvic Organ Prolapse/Incontinence Sexual Questionnaire IUGA-Revised (PISQ-IR)--Sexually Active, Assessment of Desire
Description: as for outcome 18
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Domain is relevant only the sexually active participants
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 57 | 61
units on a scale | 0.08 [-2.79 to 2.95] | -1.3 [-4.09 to 1.5]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.495, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, with unstructured variance co-variance matrix; Model based LS mean difference = -1.37, 95% CI 2-sided [-5.36 to 2.61]

27. Secondary Outcome: Change From Baseline in Pelvic Organ Prolapse/Incontinence Sexual Questionnaire IUGA-Revised (PISQ-IR)--Sexually Active, Global Quality
Description: as for outcome 18
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: Domain is relevant only the sexually active participants
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 57 | 61
units on a scale | 2.75 [-1.13 to 6.64] | -0.07 [-3.84 to 3.71]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.303, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = -2.82, 95% CI 2-sided [-8.22 to 2.59]

28. Secondary Outcome: Change From Baseline in Pelvic Organ Prolapse/Incontinence Sexual Questionnaire IUGA-Revised (PISQ-IR)--Sexually Active Interest, Assessment of Partner Related Impacts (Winsorized)
Description: Change was calculated as the followup value minus the baseline value. Change values were Winsorized at the 1st and 99th percentile. Values are model generated Least Square Means for combined 6 and 12 week time points Range of 0-100, higher score indicates better quality of life
Time Frame: Repeated change from baseline to 6 and 12 weeks
Population: as for outcome 23
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga Practice Program | Physical Conditioning Program
Number analyzed (Participants) | 50 | 50
units on a scale | -2.52 [-5.73 to 0.7] | 0.45 [-2.77 to 3.68]
Statistical Analysis 1: Comparison: Yoga Practice Program vs Physical Conditioning Program; Test type: Superiority; p = 0.196, Mixed Models Analysis; adjusted for baseline value Repeated measures mixed models, unstructured variance co-variance matrix; Model based LS mean difference = 2.97, 95% CI 2-sided [-1.56 to 7.51]

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Yoga Practice Program | Physical Conditioning Program
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/119
Serious Adverse Events (participants affected / at risk) | 1/121 | 1/119
Other Adverse Events (participants affected / at risk) | 37/121 | 43/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga Practice Program (N=121) | Physical Conditioning Program (N=119)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
High Grade B-Cell Lymphoma Burkitt-Like Lymphoma Nos (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga Practice Program (N=121) | Physical Conditioning Program (N=119)
Recurrent Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Detached Retina (Eye disorders) | 0 (0) | 1 (1)
Abdominal Cramps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 2 (2) | 2 (2)
Tooth Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Facial Pain (General disorders) | 0 (0) | 1 (1)
Allergy (Immune system disorders) | 1 (1) | 0 (0)
Allergy Nos (Immune system disorders) | 0 (0) | 1 (1)
Hay Fever (Immune system disorders) | 1 (1) | 0 (0)
Bladder Infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Coronavirus Infection (Infections and infestations) | 1 (1) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0)
Lower Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Mumps (Infections and infestations) | 1 (1) | 0 (0)
Shingles (Infections and infestations) | 1 (1) | 1 (1)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 4 (4) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Back Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Knee Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lateral Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Leg Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulled Hamstring (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shoulder Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toe Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaccination Adverse Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colonoscopy (Investigations) | 1 (1) | 0 (0)
Endoscopy (Investigations) | 0 (0) | 1 (1)
Back Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Back Pain; Knee Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Frozen Shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hand Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hip Arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hip Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Knee Swelling (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Lumbar Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain Ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Elbow (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Patellofemoral Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator Cuff Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shoulder Deformity Nos (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Shoulder Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Disorder Nos (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervical Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Localised Numbness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine, Unspecified (Nervous system disorders) | 1 (1) | 0 (0)
Neck Numbness (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica Aggravated (Nervous system disorders) | 1 (1) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma Aggravated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthmatic Attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cyst Epidermal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neck Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Back Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder Sling Procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Bunionectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee Arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Oral Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Shoulder Replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Hot Flashes (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT03672461/Prot_SAP_000.pdf